CLINICAL TRIAL: NCT05693402
Title: Efficacy of Opioid-Free Anesthesia in Modified Radical Mastectomy
Brief Title: Opioid-Free Anesthesia in Modified Radical Mastectomy
Status: Completed | Type: Observational
Sponsor: Etienne El Helou (Other)
Responsible Party: Sponsor-Investigator, Etienne El Helou, Principal investigator, Dr Etienne El Helou
Organization: Dr Etienne El Helou (Other)
Other Study IDs: HelouAssaf
Record Dates: First submitted 2022-12-16; First posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Surgery; Anesthesia; Opioid Use

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 consisting of treated patients using OFA: Group 1 consisted of 56 (Mean age was 54±14 years)
- Group 2 consisting of treated patients using NOFA: Group 2 consisted of 60 patients (Mean age was 51±12 years)
  Interventions: Procedure: opioid anesthesia

INTERVENTIONS:
Procedure: opioid anesthesia — opioid-free general anesthesia vs non opioid-free general anesthesia
  Groups: Group 2 consisting of treated patients using NOFA

SUMMARY:
The aim of this study is to evaluate the efficacy of opioid-free general anesthesia for breast surgeries in female patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwenting modified radical mastectomy
* Undergoing general anesthesia

Exclusion Criteria:

* Patients were excluded if they had Alzheimer's Disease, mental retardation, failure of locoregional anesthesia, contraindication for locoregional anesthesia.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Between January 2018 and September 2020, data from admitted patients for modified radical mastectomy under general anesthesia were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Post operative Morphone use | up to 24 hours
  Patients who received Morphine at different time points in function of the two study groups
Time To Extubation (TTE) | Directly intraOp
  Time to Extubation in function of the two study groups

SECONDARY OUTCOMES:
Post Operative Nausea and Vomiting (PONV) | Up to 24hours
  Patients who had PONV at different times in function of the two study groups

CONTACTS AND LOCATIONS:
Locations (1):
- Lebanese Hospital Geitaoui-University Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No